CLINICAL TRIAL: NCT02315313
Title: The Link Between the Clinical Resting Heart Rate and Sympathetic Overactivation
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Wang Jiguang, Director, The Shanghai Institute of Hypertension, Ruijin Hospital
Other Study IDs: ESR-14-10153
Record Dates: First submitted 2014-12-02; First posted 2014-12-11 (Estimated); Last update posted 2014-12-11 (Estimated); Status verified 2014-12

CONDITIONS: Cardiovascular Disease
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- group1: RHR≤60bpm
- group2: RHR 61-70bpm
- group3: RHR 71-80bpm
- group4: RHR >80bpm

SUMMARY:
It is a retrospective study with no products limitation to investigate the link between clinical resting HR and SOA. Use HR≤60bpm as control group, compare other three groups with the control group and find out the correlation between HR and SOA indexes.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of subject informed written or oral consent
2. Female and male aged≥ 20 to ≤ 80 years;
3. Records on mean clinical heart rate and SOA indexes were available.

Exclusion Criteria:

1. Participation in another clinical study with an investigational product during the last 6 months;
2. Drug intervention on heart rate 1 month prior to the inclusion;
3. Patients with missing data in the database from the Shanghai Institute of Hypertension, Ruijin Hospital, Shanghai.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: cardiovascular disease patient
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2014-12; Primary Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
The difference of HRV, BPV, LF/HF between each groups | 1min HR measure
  The difference on mean sympathetic overactivation related indexes such as HRV, BPV, LF/HF between groups